CLINICAL TRIAL: NCT03466008
Title: Whole-Body Cryotherapy (WBC) as an Adjunct Treatment on Pain in Fibromyalgia Persons: Short Time Effect.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haute École Robert Schuman Libramont (Other)
Responsible Party: Principal Investigator, François Tubez, Physical Therapist, PT, PhD Student, Principal investigator, Haute École Robert Schuman Libramont
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: B039201629783
Record Dates: First submitted 2018-02-02; First posted 2018-03-15 (Actual); Last update posted 2018-03-15 (Actual); Status verified 2018-03

CONDITIONS: Fibromyalgia
Keywords: whole body cryotherapy; fibromyalgia; chronic pain; quality of life; perceived health
MeSH Terms: conditions — Fibromyalgia; Chronic Pain

STUDY DESIGN:
Intervention Model Description: between (two groups: WBC and control), and within subjects (two repeated measures: pre and post intervention)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Whole body cryotherapy arm (Experimental): intervention consisted of 10 sessions of WBC (three minutes for each session) which were performed in addition to usual care in a standard cryotherapy room over a duration of 8 days.
  Interventions: Behavioral: Whole-Body Cryotherapy
- Usual treatment arm (No Intervention): usual care

INTERVENTIONS:
Behavioral: Whole-Body Cryotherapy — 10 sessions of WBC were performed (in addition to usual care) in a standard cryotherapy room over a duration of 8 days.
  Other Names: Usual intervention
  Arms: Whole body cryotherapy arm

SUMMARY:
Our aim was to determine whether Whole Body Cryotherapy (WBC) can result in improved pain status, perceived health, and quality of life in patients with fibromyalgia. It is hypothesized that this positive effect can be achieved through increased functional mobility and decreased pain intensity resulting from cold-induced modulation of the inflammation-immune axis.

DETAILED DESCRIPTION:
24 patients with fibromyalgia were randomized into 2 groups (n=11 in the WBC group, n=13 in the control group). In the WBC group, 10 sessions of WBC were performed (in addition to usual care) in a standard cryotherapy room over a duration of 8 days. Patients in the control group did not change anything in their everyday activities. Several self-reported variables relating to perceived health were measured repeatedly (pain intensity, functional mobility, and quality of life).

ELIGIBILITY:
Inclusion Criteria:

Fibromyalgia diagnosis

Exclusion Criteria:

cardiorespiratory disorder current pregnancy cold intolerance Embolic diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-04-01 (Actual); Study Completion 2017-05-30 (Actual)

PRIMARY OUTCOMES:
pain status at 1 month from baseline | change from baseline at one month follow-ups
  pain score on a numerical scale (Subjective Numerical scale) likert rating 0 to 10 by the fibromyalgia patient 0 indicate no pain, 10 maximal pain value

SECONDARY OUTCOMES:
pain status at 2 weeks from baseline | change from baseline at two weeks follow-ups
  pain score on a Subjective Numerical scale 0 to 10; likert rating 0 to 10 by the fibromyalgia patient 0 indicate no pain, 10 maximal pain value
functional status : the Oswestry Disability Index (ODI), subjective low back pain questionnaire | chnage from baseline at two weeks follow-ups
  Patient-completed questionnaire which gives a subjective percentage score of level of function (disability) in activities of daily living in those rehabilitating from low back pain There are 10 questions (items). The questions are designed in a way that to realize how the back or leg pain is affecting the patient's ability to manage in everyday life.
  Each of the 10 items is scored from 0 - 5. The maximum score is therefore 50. The obtained score can be multiplied by 2 to produce a percentage score.
  If the first statement is marked, the section score = 0, If the last statement is marked, it = 5
  If all ten sections are completed the score is calculated as followed:
  Example: 10 (total score of the patient), 50 (total possible raw score), 10/50 x 100 = 20%
  If one section is missed or not applicable, the score is calculated as followed:
  Example: 15 (total score of the patient), 45 (total possible score), 15/45 x 100 = 30%
functional status : the Oswestry Disability Index (ODI) | change from baseline at one month follow-ups
  Patient-completed questionnaire which gives a subjective percentage score of level of function (disability) in activities of daily living in those rehabilitating from low back pain There are 10 questions (items). The questions are designed in a way that to realize how the back or leg pain is affecting the patient's ability to manage in everyday life.
  Each of the 10 items is scored from 0 - 5. The maximum score is therefore 50. The obtained score can be multiplied by 2 to produce a percentage score.
  If the first statement is marked, the section score = 0, If the last statement is marked, it = 5
  If all ten sections are completed the score is calculated as followed:
  Example: 10 (total score of the patient), 50 (total possible raw score), 10/50 x 100 = 20%
  If one section is missed or not applicable, the score is calculated as followed:
  Example: 15 (total score of the patient), 45 (total possible score), 15/45 x 100 = 30%
functional status : the Disability of the Arm, Shoulder and Hand (DASH) score | change from baseline at one month follow-ups
  The Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire is a 30-item questionnaire that looks at the ability of a patient to perform certain upper extremity activities. This questionnaire is a self-report questionnaire that patients can rate difficulty and interference with daily life on a 5 point Likert scale. DASH Scoring Formula = ([(sum of n responses)/n] -1)(25) where n represents the number of completed items. The score on both test ranges from 0 (no disability) to 100 (most severe disability).Minimal Detectable Change (MDC) is between 12.75% - 17.23%
functional status : Lower Extremity Functional Scale (LEFS) | change from baseline at one month follow-ups
  The test can be used to evaluate the impairment of a patient with lower extremity musculoskeletal condition or disorders. Can be used clinically to measure the patients' initial function, ongoing progress, and outcome as well as to set functional goals.In 1999, Binkley et al. developed the Lower Extremity Functional Scale (LEFS), a patient-reported lower limb function questionnaire applicable to a wide spectrum of outpatients with a lower limb musculoskeletal condition. The LEFS consists of 20 items, each scored on a 5-point scale (0 to 4). The total score varies from 0 to 80, with higher scores representing better a functional status.
health related quality of life (HRQoL) | change from baseline to one month follow-ups
  physical functioning (PCS) and mental functioning (MCS) from the SF-36 questionnaire The score on both test ranges from 0 (poor health related quality of life) to 100 (better health related quality of life value)

CONTACTS AND LOCATIONS:
Overall Officials: guillaume polidori, Pr, Study Director — University of Reims

IPD SHARING:
Plan to Share IPD: No
confidential personal data